CLINICAL TRIAL: NCT01692158
Title: Pharmacodynamics Study of Enoxalow, Produced by Blau Farmacêutica S/A, Compared to Clexane, Produced by Sanofi-Aventis Farmacêutica Ltda, in Healthy Subjects After Subcutaneous Administration.
Brief Title: Pharmacodynamics Study of Enoxalow Compared to Clexane in Healthy Subjects After Subcutaneous Single Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ENOBLA0512SC-I; Versão 01 datada de 15.05.2012 (Other: LAL Clinica)
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Healthy
Keywords: subjects
MeSH Terms: interventions — Heparin, Low-Molecular-Weight; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teste (Experimental): Enoxalow (Heparin, Low-Molecular-Weight) - Blau Farmacêutica S/A.
  Interventions: Drug: Heparin, Low-Molecular-Weight
- Comparador (Active Comparator): Clexane (Heparin, Low-Molecular-Weight)- Sanofi-Aventis
  Interventions: Drug: Heparin, Low-Molecular-Weight

INTERVENTIONS:
Drug: Heparin, Low-Molecular-Weight — single subcutaneuous administration of 40 mg of the test drug and the comparator drug, according to randomization, in a crossover design, each administration separated by 6 days of washout.
  Other Names: Clexane; Enoxalow

SUMMARY:
The hypothesis of this trial is that the test drug (Enoxalow® - T) pharmacodynamics parameters are similar to the comparator drug (Clexane® - C) in healthy subjects following administration of single subcutaneous dose. The objective of this randomized, crossover, clinical trial is to evaluate the pharmacodynamic profile of the test drug Enoxalow® - T produced by Blau Farmacêutica, compared to the comparator drug Clexane®, produced by Sanofi-Aventis, by determining pharmacodynamic activities (including anti FXa and anti-FIIa), as surrogate markers for their circulating concentrations of the drug.

DETAILED DESCRIPTION:
In addition other pharmacodynamic tests such as Tissue Factor Pathway Inhibitor (TFPI) activity, as well as the ratio of anti-FXa and anti-FIIa activity will be compared as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Agree to all the purposes of the study by signing and dating the Informed Consent;
* Male, aged between 18 and 55 years, clinically healthy;
* BMI between 18.5 and 30;

Exclusion Criteria:

* Participation in clinical trials in the 12 months preceding the trial;
* Presence of pulmonary, cardiovascular, neurological, endocrine, gastrointestinal, genitourinary or other systems diseases;
* Acute disease in the period of 07 days before the beginning of the practical phase (administration of the drug) of the study;
* Chronic administration of medications for hypertension, diabetes or any other disease that requires continuous use of any drug;
* Hemoglobin < 13 g/dL;
* Continuous use of oral anticoagulants, platelet inhibitors or anti-inflammatory drugs;
* Use of medications that interact with enoxaparin;
* History of gastrointestinal bleeding, deep vein thrombosis or pulmonary embolism that may interfere with the clinical outcome of the study;
* History of coagulopathy and bleeding diathesis;
* Presence of changes in physical examination suggestive of coagulation disorders (bruising, petechiae, or bruising);
* Changes in the skin or subcutaneous tissue of the place of drug administration(eg liposuction in the abdomen);
* Absolute platelet count below 100 x 109 / L;
* History of chronic bleeding;
* History of acute haemorrhage in the past 30 days;
* History of sensitivity to mammalian-derived biological products, albumin or any component of the formulation;
* History of allergy or Steven Johnson disease;
* Current or previous history (under 12 months) use of illicit drugs and tobacco;
* History of alcohol abuse, current or previous (within 12 months);
* At the discretion of the Principal Investigator of the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
anti-FXa | 0, 0:30, 1, 1:30, 2, 2:30, 3, 3:30, 4, 4:30, 5, 6, 8, 10, 12, 16, 20 and 24h after drug administration
anti-FIIa activity | 0, 0:30, 1, 1:30, 2, 2:30, 3, 3:30, 4, 4:30, 5, 6, 8, 10, 12, 16, 20 and 24 hours after drug administration

SECONDARY OUTCOMES:
Tissue Factor Pathway Inhibitor (TFPI) | 0, 0:30, 1, 1:30, 2, 2:30, 3, 3:30, 4, 4:30, 5, 6, 8, 10, 12, 16, 20 and 24 hours after drug administration
ratio of anti-FXa and anti-FIIa activity | 0, 0:30, 1, 1:30, 2, 2:30, 3, 3:30, 4, 4:30, 5, 6, 8, 10, 12, 16, 20 and 24h after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Frederico, Principal Investigator — Azidus Brasil
Locations (1):
- LAL Clinica, Valinhos, São Paulo, Brazil